CLINICAL TRIAL: NCT05324631
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase 3 Clinical Study to Evaluate the Efficacy and Safety of SHR0302 in Active Non-Radiographic Axial Spondyloarthritis Subjects
Brief Title: A Study to Evaluate the Efficacy and Safety of SHR0302 in Patients With Non-Radiographic Axial Spondyloarthritis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHR0302-305
Record Dates: First submitted 2022-04-06; First posted 2022-04-12 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Non-radiographic Axial Spondyloarthritis
MeSH Terms: conditions — Non-Radiographic Axial Spondyloarthritis | interventions — ivarmacitinib

STUDY DESIGN:
Intervention Model Description: SHR0302 compared with placebo
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental): SHR0302
  Interventions: Drug: SHR0302
- Treatment group B (Placebo Comparator): SHR0302 Placebo
  Interventions: Drug: SHR0302 placebo

INTERVENTIONS:
Drug: SHR0302 — SHR0302, oral, once daily
  Arms: Treatment group A
Drug: SHR0302 placebo — SHR0302 placebo, oral, once daily
  Arms: Treatment group B

SUMMARY:
This study is to evaluate the efficacy and safety of SHR0302 in subjects with active non-radiographic axial spondyloarthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed informed consent.
2. BMI ≥18 kg/m2.
3. Participant has the clinical diagnosis of nr-axSpA fulfilling the 2009 ASAS classification criteria for axSpA but not meeting the radiologic criterion of the modified New York criteria for AS and have objective signs of active inflammation on magnetic resonance imaging (MRI) or based on high sensitivity C-reactive protein (CRP).
4. Participant must have baseline disease activity as defined by having a Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score >= 4 and a Patient's Assessment of Total Back Pain score >= 4 based on a 0 - 10 Numeric Rating Scale (NRS) at the Screening and Baseline Visits.
5. Participant has had an inadequate response to at least two Nonsteroidal Anti-inflammatory Drugs (NSAIDs) over an at least 4-week period in total at maximum recommended or tolerated doses, or participant has an intolerance to or contraindication for NSAIDs as defined by the Investigator.
6. If subjects are taking permitted csDMARDs or low-dose corticosteroid orally at baseline, the stable doses should have lasted for more than 4 weeks already.

Exclusion Criteria:

1. Pregnant women or refuse to receive contraception during the study.
2. Lab abnormality within 4 weeks of randomization as follows: WBC count <3.0×10^9/L；neutrophil count<1.5×10^9/L;hemoglobin level<90.0 g/L ; platelet count <100×10^9/L; AST or ALT levels greater than the 1.5 times the upper limit of normal; HBsAg or HCV or HIV antibody positivity.
3. History of other autoimmune diseases ; history of cancer or infection including tuberculosis and hepatitis; history of important cardiovascular events or thrombotic diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-08-16 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-12-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Assessment of SpondyloArthritis International Society (ASAS) 40 Response at week 12 | Week 12

SECONDARY OUTCOMES:
Change From Baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS) at week 12 | Week 12
Percentage of Participants With ASAS 20 Response at week 12 | Week 12
Change from baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at week 12 | Week 12
Percentage of Participants with ASAS 5/6 response at Week 12 and Week 24 | Week 12 and Week 24
Change from baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) at Week 12 and Week 24 | Week 12 and Week 24
Change from baseline in Bath Ankylosing Spondylitis Metrology Index (BASMI) at Week 12 and Week 24 | Week 12 and Week 24
Change from baseline in Short-Form-36-Health Survey (SF-36) at Week 12 and Week 24 | Week 12 and Week 24
Change from baseline in Ankylosing Spondylitis Quality of Life (ASQoL) at Week 12 and Week 24 | Week 12 and Week 24

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided